### IND #112478, STUDY PROTOCOL 3 **UW/FHCRC Cancer Consortium IRB # 7754**

TITLE:

Cellular Proliferation Imaging Using [18F] fluorothymidine (FLT)

Positron Emission Tomography (PET) in Brain Tumors

Principal Investigator:

Jason K. Rockhill, M.D. Ph.D.

University of Washington Medical Center

1959 NE Pacific St.,

Box 356043

Seattle, Washington 98195 Telephone: (206) 598-4121 Fax: (206) 598-3786 jrock@u.washington.edu

Sub-Investigators:

Janet F. Eary, MD

Department of Radiology University of Alabama

JT N412

619 19th St South

Birmingham AL 35249-6830 Phone: 205-934-3138 jeary@uabmc.edu

James R. Fink, M.D.

University of Washington Medical Center

1959 NE Pacific St., Rm NW011

Box 357115

Seattle, WA 98195

Telephone: (206) 543-3320

Fax: (206) 598-8475 jrfink@u.washington.edu

Daniel L. Silbergeld, M.D.

University of Washington Medical Center 1959 NE Pacific St., Rm. RR744-C

Box 356470

Seattle, WA 98195

Telephone: (206) 543-3570

Fax: (206) 543-8315

dls@u.washington.edu

FHCRC IRB Approval

OCT 26 2016

Robert C. Rostomily, M.D.

University of Washington Medical Center

1959 NE Pacific St., Rm. RR744

Box 356470

Seattle, WA 98195

Telephone: (206) 543-3570, 543-8043

Fax: (206) 543-8315 rosto@u.washington.edu Document Released Date

Maciej M. Mrugala, M.D., Ph.D. University of Washington Medical Center 1959 NE Pacific St. Box 356097 Seattle, WA 98195 Telephone: (206) 598-9487 Fax: (206) 598-7919 mmrugala@u.washington.edu

Lia Halasz, M.D.
University of Washington Medical Center
1959 NE Pacific St.
Box 356043
Seattle, WA 98195
Telephone: (206) 598-4100
Fax: (206) 598-3786
Ihalasz@u.washington.edu

Manuel Ferriera
University of Washington Medical Center
1959 NE Pacific St.
Box 356470
Seattle, WA 98195
Telephone: (206) 543-3570
Fax: (206) 543-8315
manuelf3@u.washington.edu

Andrew Shields, M.D.
University of Washington Medical Center
1959 NE Pacific St., Rm NW041
Box 356113
Seattle, WA 98195-6004
Telephone: (206) 559-6856
Fax: (206) 598-4192
andrews@u.washington.edu

Jean H. Lee, M.D.
University of Washington Medical Center
1959 NE Pacific St. Rm. BB308
Box 357115
Seattle, WA 98195-6004
Telephone: (206) 598-0024
Fax: (206) 598-0252
jeanhlee@u.washington.edu

Kenneth A. Krohn, Ph.D. University of Washington Medical Center 1959 NE Pacific St., Rm NW055 Box 356004

Seattle, WA 98195-6004 Telephone: (206) 598-6245 Fax: (206) 598-4192

kkrohn@u.washington.edu

Dr. Krohn is a radiochemist and is not involved in patient care

Jeanne M. Link, Ph.D.
Oregon Health Sciences and University
3181 SW Sam Jackson Park Road
Mail Code L340
Portland, OR 97239
Telephone: (206) 406-4509
Fax: (503) 494-4982

Fax: (503) 494-4982 lijea@ohsu.edu

Dr. Link is a radiochemist and is not involved in patient care.

Steven C. Shoner, PhD University of Washington Medical Center Box 356004 Seattle, WA 98195-6004 Telephone: (206) 598-6711 Fax: (206) 598-4192

scshoner@u.washiongton.edu

Dr. Shoner is a radiochemist and is not involved in patient care.

## Study Coordinator / Data Managers:

Kristin Kauno, CCRC
University of Washington Medical Center
1959 NE Pacific St., Rm NW041
Box 356004
Seattle, WA 98195-6004
Telephone: (206) 598-7883
Fax: (206) 598-7540
kkauno@u.washington.edu

Mark Muzi, M.S.
University of Washington Medical Center
1959 NE Pacific St., HSB NW-134B
Box 356004
Seattle, WA 98195-6004
Telephone: (206) 543-3517
Fax: (206) 685-6473

Fax: (206) 685-6473 muzi@u.washington.edu **Statistical Consultant** 

Finbarr O'Sullivan, Ph.D.

University College Cork

School of Mathematical Sciences

Room 1-57 first floor

Western Gateway Building, Western Road

Cork, Ireland

Telephone: 011-353-214-902826 Fax: 011-353-214-4295364

f.osullivan@ucc.ie

Dr. O'Sullivan is a statistician and is not involved in patient care.

**Current Version Number: 7** 

**Current Protocol Version Date:** 03/08/2016 **Previous Protocol Version Date:** 12/12/14

# TABLE OF CONTENTS Protocol 3: Cellular Proliferation Using [18F]-Fluorothymidine(FLT) Positron Emission Tomography (PET/CT) in Brain Tumors

| | | Page |
|---|---|---|
| 6.iii.1. Sch | nema | 6 |
| 6.iii.2. Obj | ectives | . 7 |
| 6.iii.2.a. | Specific Aims | . 7 |
| 6.iii.3. Bad | ckground | 7 |
| | Study Disease | |
| | Investigational Agent | |
| | Rationale | |
| 6.iii 4 Pat | tient Selection | 10 |
| | Inclusion Criteria | |
| | Exclusion Criteria. | |
| | Inclusion of Women and Minorities | |
| | Accrual Targets | |
| 6.iii.5. Reg | gistration Procedures | . 12 |
| 6.iii.6. Tre | eatment Plan | . 12 |
| | [ <sup>18</sup> F]FLT Administration | |
| | Study Procedures and Schedule of Events | |
| | General Concomitant Medication and Supportive Care Guides | |
| | Duration of Therapy | |
| | Duration of Follow Up | |
| 6.iii.7. Exp | pected Toxicities and Dosing Delays / Dose Modifications | . 14 |
| Aiii A Ad | verse Events Reporting | 1/ |
| | General Definitions. | |
| | Adverse Events Reporting Requirements | |
| | CAEPR / ASAE for [18F]FLT. | |
| | Potential but Unexpected AEs for [18F]FLT | |
| | Review of Safety Information | |
| | Adverse Event Reporting | |
| | Expedited Adverse Reaction Reporting Guidelines | |
| | Protocol-specific Expedited AE Reporting Exclusion | |
| | Routine Adverse Event Reporting | |
| 6.iii.9. Pha | armaceutical Information | . 19 |
| 6.iii.9.a. | Production of Radiopharmaceutical | . 19 |
| 6.iii.9.b. | Reported Adverse Events and Potential Risks | 19 |
| | Agent Accountability | |

| 6.iii.10. Correlative Studies | 20 |
|------------------------------------------------------|----|
| 6.iii.10.a. [18F]FLT PET/CT Image Analysis | |
| 6.iii.10.b. Biologic Correlates | 21 |
| 6.iii.11. Study Calendar | 21 |
| 6.iii.12. Measurement of Effect | 21 |
| o.iii. 12. Measurement of Effect | 21 |
| 6.iii.13. Data Reporting / Regulatory Considerations | 23 |
| 6.iii.14. Statistical Consideration | 23 |
| 6.iii.14.a Study Description | |
| 6.iii.14.b Power Calculations | |
| 6.iii.14.c Analysis Plan | |
| 6.iii.14.d Stratification Factors | 25 |
| 6.iii.14.e Reporting and Exclusions | |

### 6.iii.1. SCHEMA

This clinical study will obtain preliminary data to investigate the role of [18F]FLT in patients with primary or recurrent brain tumors that will be undergoing tumor therapy. This study will obtain data on the value of [18F]FLT to quantify uptake changes related to cellular proliferation using serial scans, which will include a baseline scan prior to therapy, and follow-up scans after standard therapy has started. If promising, these data will be used to design larger clinical trials.

Cellular proliferation imaging with specific PET agents provides a unique approach to quantify the growth rate of tumors and assess their treatment response. Our research group pioneered the development and validation of [18F]fluorothymidine (FLT) as a tracer of cellular proliferation. FLT has been shown to accumulate in tissues in proportion to the level of *thymidine kinase I* activity. This enzyme is up-regulated during the DNA synthesis portion of the cell cycle and therefore its activity reflects cellular proliferation. We will use this FLT biochemical marker using PET/CT to quantify regional cellular growth rate in brain tumors. These tumors are known to have high levels of proliferation, which can change with treatment. Our hypothesis is that quantifying cellular proliferation in brain tumors will provide a useful measure of disease activity and location.

# STUDY PROTOCOL SEQUENCE Clinical diagnosis of a brain tumor eligible for therapy Study Registration Pre-Therapy FLT PET/CT Scan 1 (DYNAMIC 1 field of view) Blood collection for metabolite analysis Mid-therapy FLT PET/CT Scan 2 (DYNAMIC 1 field of view) Blood collection for metabolite analysis Completion of therapy or clinical follow-up FLT PET/CT Scan 3 and at recurrence potential Scan 4 (DYNAMIC 1 field of view) Blood collection for metabolite analysis Clinical Follow up as long as the patient is seen in UW clinics. Standard adjuvant therapy as directed by treating clinician. Additional imaging (MR) as clinically indicated.

Figure 6.iii.1. Schema for brain tumor protocol

We emphasize that this is an observational study in that [18F]FLT PET/CT will not be used to direct therapy. Treatment regimens are chosen by the referring oncologist prior to the [18F]FLT PET study on the basis of clinical criteria. While patients and referring physicians will not be blinded to [18F]FLT PET results, treatment choices will be made prior to the entry of the patient into the study and clinical management will be based on usual standard-of-care anatomic MRI and/or FDG PET/CT and will not be altered because of the FLT PET/CT results.

### 6.iii.2. OBJECTIVES

### 6.iii.2.a. Specific Aims:

- 6.iii.2.a.1. Using FLT PET/CT as a measure of cellular proliferation, assess tissue proliferation in disease sites of brain tumor patients before therapy (surgery, chemotherapy or radiotherapy or any combination of these.).
- 6.iii.2.a.2. Determine level of change in cellular proliferation compared with baseline (Scan 1) in brain tumors at mid-therapy (Scan 2), after completion of therapy (Scan 3) and in the clinical follow-up period (Scan 4), when possible.
- 6.iii.2.a.3. Correlate levels of cellular proliferation measured by FLT PET/CT at baseline and treatment-induced changes in brain tumor proliferation with clinical response status (clinical categories are complete remission, lesser degrees of response/stable disease, and no response).
- 6.iii.2.a.4. Assess spatial heterogeneity of FLT uptake to identify local differences in brain tumor disease burden. This aim is a secondary analysis. For patients in which re-operation is clinically indicated, we will mark surgical specimens to co-register with regions of the FLT image. These tissues will be banked for future histological assays.

### 6.iii.3. BACKGROUND

Cellular proliferation imaging with specific PET agents provides a noninvasive approach to quantify the growth rate of tumors serially and to assess their treatment response. Our research group pioneered the development and validation of [18F]-fluorothymidine (FLT), which has been shown to accumulate in tissues in proportion to the level of cellular growth (Shields, 1998; Krohn, 2012). During cellular uptake, FLT is transported across the cell membrane and then phosphorylated by *thymidine kinase-1*, resulting in intracellular trapping of the radiolabeled nucleotide (Grierson, 2004). Because of the substitution at the 3'-position, FLT is not a good substrate for *DNA polymerase*. *Thymidine kinase-1* activity is controlled throughout the cell cycle processes, which forms the basis for relating FLT uptake to cellular proliferation. Although FLT is not incorporated into DNA, its retention in cells is directly related to *thymidine kinase-1* activity, which peaks in S-phase and then is destroyed as the cells proceed to division (Weber, 1991; Eriksson, 1994). Our research has shown that uptake is also influenced by blood flow, which led us to develop a simple dynamic PET imaging method to obtain quantitative tissue proliferation rate information separate from tumor blood flow (Muzi


2006, Wells 2002a). PET has the ability to image the whole body and yield quantitative regional tissue information on a specific biological process. We will exploit this approach in this study of FLT PET/CT to quantify regional cellular growth rate in primary brain tumors.

### 6.iii.3.a. Study Disease

Brain tumors: Brain tumors are known to have variable levels of cellular proliferation which is also thought to be heterogeneous in the tumor volume. These tumor characteristics may be very important factors in treatment resistance. Our hypothesis is that quantifying cellular proliferation in brain tumors will provide a useful measure of disease activity. The brain malignancies are a group of tumors where dramatic responses with long-term survival can occur, but also where many patients' exhibit treatment resistance and have very short survival.

Standard initial treatment for glioblastoma currently consists of surgical removal of as much of the MRI contrast-enhancing lesion as can be accomplished safely, followed by radiotherapy and temozolomide (TMZ) chemotherapy for 6 weeks. Unfortunately, early treatment failures occur in 30-50% of patients. This definition of treatment failure is described as an increase in the MRI T1+Gd tumor volume (de Wit, 2004). Immediate post-radiotherapy MRI changes in malignant glioma can mimic tumor progression (Taal, 2008). The incidence of this pseudo-progression in a cohort of malignant glioma patients treated with chemo-radiation with temozolomide is significant (Brandes, 2008). From 28-52% of these patients will demonstrate improvement on subsequent MRI studies when they continue on standard TMZ chemotherapy. This situation defines pseudoprogression as opposed to true disease progression, where continued treatment with temozolomide is associated with continued clinical decline and MRI T1+Gd worsening. Clinicians armed with anatomic MRI imaging alone may wrongly conclude that standard treatment is failing in these patients, leading to cessation of a treatment that is actually working. Also, misdiagnosing pseudo-progression in patients who are responding could risk entering such patients into phase II or III trials of new agents, decreasing the statistical power of the study and potentially leading to falsely positive outcomes. On the other hand, continuing TMZ in the patients that are true progressors wastes their time and physiological resources when they should be offered second line treatment or enrollment in a phase II or III research treatment protocol. Thus, the ability to make the important distinction between progression and pseudo-progression is critical for the care of treated brain tumor patients and could potentially change patient management. In some patients, the neuropathologist who reviews the resected tumor resolves the question of pseudo-progression versus true progression. Ideally, however, noninvasive imaging methods should be developed to answer this question reliably. Our primary hypothesis is that FLT PET/CT should be able to distinguish between when the patient has true tumor progression and needs to change therapy and when the MRI contrast is reflecting pseudo-progression and the patient should continue with TMZ chemotherapy. That way, the 50% or possibly more true progressors could avoid continuing futile TMZ.

Recent reviews have described many alternative strategies for overcoming treatment resistance for therapy with new combination protocols. One example is the addition of bevacizumab to the TMZ-radiotherapy combination to normalize vascular permeability changes at the time of radiologic signs of pseudo-progression, but the change in patient outcome for this therapy addition is unknown (Villano, 2009). Increases in radiotherapy


with stereotactic and brachytherapy techniques are also showing results with cautious increases in treatment dose, and little increased toxicity (Fokas, 2009, Fabrini, 2009). Other attempts at tumor re-resection in patients with recurrent tumors or progression is historically shown to be effective for only a subset of patients, leading to exploration of the clinical utility of drugs designed to target specific tumor mechanisms for cell growth and maintenance. However, many of these targeted agents have not demonstrated improved survival in groups of non-selected patients (Sathornsumetee, 2009). While MR methods in aggregate may have the ability to distinguish true treatment responses prospectively, there is little agreement on techniques to apply consistently to make this critical clinical diagnosis in an individual patient. The new research of this study will evaluate PET approaches to these important clinical questions. If FLT PET/CT can accurately identify true progression, then this imaging protocol can be used for following response to current therapy and for objective evaluation of the promise of newer molecularly targeted therapies for patients with malignant brain tumors. Tumor proliferation imaging will enable us to observe the location and distribution of disease throughout the course of treatment to gain new insight into a patient's progress and about brain tumor biology. The goal of this project is to provide objective and quantitative imaging information about the entire brain tumor in a pilot study that builds on our substantial work in FLT-PET applied to human cancer.

### 6.iii.3.b. Investigational Agent

3'-Deoxy-3'-[<sup>18</sup>F]fluorothymidine ([<sup>18</sup>F]FLT) is a structural analog of the DNA constituent, thymidine (Figure 6.iii.2). It is a radiolabeled imaging agent that has been proposed for investigating cellular proliferation with positron emission tomography (PET). Although [<sup>18</sup>F]FLT is not incorporated into DNA, it is trapped in the cell due to phosphorylation by thymidine kinase 1, a part of the salvage pathway. As such, it has potential as a marker of proliferating tumor in proportion to the DNA synthesis rate. Therefore, [<sup>18</sup>F]FLT is proposed as a radiolabeled imaging probe for *in vivo* assessment of cellular proliferation in malignant tumors using PET. For complete information, please refer to the Investigator's Brochure: "3'-deoxy-3'-fluorothymidine: [<sup>18</sup>F]FLT, An Investigational Positron Emission Tomography (PET) Radiopharmaceutical for Injection and intended for use as an in vivo diagnostic for imaging active cellular proliferation of malignant tumors."

### 6.iii.3.c. Rationale

[18F]FLT is a radiolabeled imaging probe for *in vivo* assessment of cellular proliferation using PET. Preclinical and clinical studies suggest that early imaging of response using this radiopharmaceutical can demonstrate effectiveness of treatment in a variety of tumors. In this protocol, we will assess regional FLT uptake in patients with malignant brain tumors.

Figure 6.iii.2. Molecular structures for FLT and thymidine

Specifically, we propose to use [18F]FLT PET/CT to assess changes in imaging measures in the clinical course of brain tumor patients. Subsequent studies (not part of this trial) could eventually allow treatments to be tailored to the tumor response measured by imaging, eliminating the use, costs and toxicity of ineffective treatments and improving the patient's quality of life. This is our long-term objective. In this protocol, FLT PET/CT imaging measures will be compared with clinical measures of tumor response to test specific hypotheses.

### Hypotheses for this protocol.

- Quantifying tumor proliferation in brain tumors will provide a reliable measure of disease. For example, kinetic analysis of the FLT-PET/CT data will allow distinction between true progression and pseudoprogression in patients with glioblastoma who have finished surgery plus radiotherapy and temozolomide and whose measurable disease by standard MRI after initial treatment has appeared to progress.
- Changes in tumor proliferation (FLT flux) as determined by kinetic analysis of FLT-PET/CT imaging will correlate with clinical treatment response.
- Brain tumor cellular proliferation is heterogeneous. This heterogeneity can be quantified by the FLT PET/CT procedure and is an independent predictor of response.

### 6.iii.4. PARTICIPANT SELECTION

### 6.iii.4.a. Inclusion Criteria:

- 6.iii.4.a.1. At least 18 years of age.
- 6.iii.4.a.2. Have a diagnosis or suspected diagnoses of a brain tumor (primary, recurrent, or metastatic) by standard clinical diagnosis such as pathology or imaging.
- 6.iii.4.a.3. Planned for treatment with radiation, chemotherapy and surgical resection or any of these treatment strategies combined. The clinical treatment will not be influenced by the experimental imaging studies described in this protocol.

### 6.iii.4.b. Exclusion Criteria:

- 6.iii.4.b.1. Inability to provide informed consent
- 6.iii.4.b.2. Pregnancy
- 6.iii.4.b.3. Inability to lie still for the imaging study
- 6.iii.4.b.4. Weight over 350 lbs., the weight limit of the tomograph table.

### 6.iii.4.c. Inclusion of Women and Minorities

Patients 18 years of age or older with a brain tumor and planning to undergo therapy will be eligible for study participation.

No other discriminatory factors, including age, sex, or ethnic background will be used to determine eligibility. Every effort will be made to ensure that minorities are recruited for study participation.

### 6.iii.4.d. Accrual Targets

Brain tumors in adults may have low incidence in some ethnic and racial groups. We have not excluded any ethnic or racial groups from participation in our studies and will continue this policy, but anticipate that some ethnic and racial groups will not enroll due to the rarity of presentation. (Table 6.iii.1) The targeted enrollment is for a total of 30 patients with three to four FLT PET/CT scans per patient. We recognize that some patients, though willing, will be too sick to be able to complete three studies which is the number required for the power calculations described in Data Analysis, section 6.iii.14.b. From our experience with this patient group, we estimate that 25% of our patients will only receive one or two scans. Therefore, we will enroll up to 40 subjects to the study. The current funding level of our NCI Program Project imposes a practical limit on the total accrual number. We fully appreciate that this will impact the statistical power. Nevertheless, because proliferation changes greatly with therapy, we are optimistic that the study will lead to significant findings on our proposed hypotheses (see Statistical Analysis, section 6.iii.14).

Table 6.iii.1. Targeted Enrollment.

| TARGETED/PLANNED ENROLLMENT: Number of Subjects (must provide actual numbers. (i.e. no range) | | | |
|---|---|---|---|
| Ethnic Category | Sex/Gender | | |
| | Females | Males | Total |
| Hispanic or Latino | 2 | 3 | 5 |
| Not Hispanic or Latino | 14 | 21 | 35 |
| Ethnic Category Total of All Subjects* | 16 | 24 | 40 |
| Racial Categories American Indian/Alaska Native | 1 | | 3 |
| Asian | <del> </del> | 1 1 | <del> </del> |
| Native Hawaiian or Other Pacific<br>Islander | 0 | 1 | 1 |
| Black or African American | 0 | 1 | 1 |
| White | 15 | 19 | 34 |
| Racial Categories: Total of All<br>Subjects | 16 | 24 | 40 |

### 6.iii.5. REGISTRATION PROCEDURES

Not applicable; this is a single institution trial.

### 6.iii.6. TREATMENT PLAN

This is not a treatment trial. Patients will be managed according to the plan developed by their treating clinicians. Patients will be treated at the University of Washington clinics where standard of care for treatment calls for surgery, chemotherapy, radiation, or chemoradiation with adjuvant chemotherapy. Standard salvage therapy will be offered patients who progress based on current clinical indications by their clinicians. Salvage therapy includes re-operation, re-irradiation, second line chemotherapy agents or a combination of these options. We will serially image patients using FLT PET/CT for quantifying tumor cellular proliferation at several time points in their clinical course. The times will include baseline and can include mid therapy and up to two scans during the clinical follow-up period after therapy. Standard clinical MR images will be acquired during the therapy schedules as requested by the clinicians. Patients may also undergo research MR imaging.

### 6.iii.6.a. [18F]FLT Administration:

[18F]FLT will be administered in the PET Imaging Suite at the University of Washington Medical Center or at the Seattle Cancer Care Alliance (SCCA). Upon arrival, the patient will have an opportunity to have questions answered regarding the procedure. The patient will have one intravenous line placed prior to [18F]FLT administration. The patient will then be positioned in the PET scanner followed by a transmission scan using a low-dose CT scan. Then [18F1FLT will be administered intravenously by a physician. The administered dose will be 0.07 mCi/kg with a maximum of 5 mCi. The drug solution is stored at room temperature in a gray butyl septum sealed, sterile, pyrogen-free glass vial and has an expiration time of 8 hours. The injectable dose of [18F]FLT will be ≤ 0.07 mCi/kg of fluorine-18, not to exceed 5 mCi. In the dose of [18F]FLT, only a small fraction of the FLT molecules are radioactive. The amount of injected drug is  $\leq 6.1 \,\mu g$  ( $\leq 25 \,nmol\,per\,dose$ ) of FLT. There is no evidence that nonradioactive and radioactive FLT molecules display different biochemical behavior. [18F]FLT is administered to subjects by intravenous injection of ≤ 10 mL. The injection will be infused over approximately 1 minute and followed by a saline flush. The infusion and imaging procedure will be terminated in any patient who exhibits anaphylaxis, significant dyspnea or chest pain.

The adverse events to be specifically monitored during the infusion include localized discomfort at the IV injection site, pain, respiratory difficulties, flushing, dizziness, pruritus/rash, and any other symptoms that could be secondary to an anaphylactic reaction. The subject will be instructed to report any subjective symptoms or sensory changes noted. All adverse events occurring post [18F]FLT infusion will be recorded within a 24-hour period.

### 6.iii.6.b. Study Procedures and Schedule of Events:

**6.iii.6.b.1. Initial visits prior to [18F]FLT PET:** Patients who are identified as potential candidates for the [18F]FLT PET study will be approached to explain the nature of the study and to obtain their written informed consent to be enrolled in the protocol. The following additional patient data will be obtained: tumor location, correlative imaging findings, histologic diagnosis (if available), age at diagnosis, and gender.

**6.iii.6.b.2. Day of [¹8F]FLT PET Scans:** The patient will be positioned supine in the PET/CT scanner for a dynamic scan over the brain. [¹8F]FLT PET/CT will be performed using the standard dose of 5 mCi. Patients will have 1 or 2 intravenous lines placed. A low-dose CT scan (PET/CT) will be used for positioning and attenuation correction. The single field of view over the brain will be imaged dynamically for about 90 minutes following the start of a one-minute intravenous infusion of [¹8F]FLT. Total patient time, including line placement and imaging is typically 2 hours. During the scan, three venous blood samples will be taken to analyze for FLT metabolites by the method we developed and is detailed in the Investigator's Brochure our previously developed solid phase exchange method that is published on the ACRIN trials website (ref: http://www.acrin.org/Portals/0/Protocols/6689/imaging/ACRIN%206689% 20FLT%20Blood%20Processing%20-

%20V1.0%20%20%20%20February%2011,%202011.pdf).

**6.iii.6.b.3.** After the baseline and follow up [<sup>18</sup>F]FLT PET Scans: A follow up phone call will be made by study staff the next day after a [<sup>18</sup>F]FLT PET/CT scan to ask about any signs of adverse effects.

### 6.iii.6.c. General Concomitant Medication and Supportive Care Guidelines

There are no requirements for concomitant medication supportive care as part of this study.

### 6.iii.6.d. Duration of Therapy:

As this is an observational study, the results of [18F]FLT PET/CT are not used to direct therapy. The duration of therapy is determined on the basis of clinical grounds by the referring physician, and is not influenced by the FLT study.

### 6.iii.6.e. Duration of Follow Up:

Patients will be followed until the time of their treatment failure or they are otherwise lost to follow-up, at which time they are considered off study. This is typically 5 years or less but may be as great as 7 years. Patients lost to follow-up will be tracked for overall survival to every extent possible based on information from public databases.

### 6.iii.7. EXPECTED TOXICITIES AND DOSING DELAYS / DOSE MODIFICATIONS

Not applicable to an observational imaging trial.

### 6.iii.8. ADVERSE EVENTS REPORTING

Qualifying Adverse Events (AEs), including Serious Adverse Events (SAEs), as defined herein, will be reported via the FDA Adverse Event Expedited Reporting System (AERS). For this IND we will report adverse events based on the FDA final rule for IND safety reporting requirements under 21 CFR part 312 published on September 29, 2010 and implemented on March 28, 2011. This investigational study is not a BA or BE study so 21 CFR part 320 is not applicable. Adverse events will also be reported to the local IRB according to their requirements.

### 6.iii.8.a. General Definitions (from 21 CFR 312.32 (a))

Adverse Event (AE): An Adverse Event is an untoward medical occurrence associated with the use of the drug in humans, whether or not considered drug related. For this study the drug is [18F]FLT and adverse events would include any events experienced by a study participant during the Adverse Event reporting period defined in Table 6.iii.4 Study Calendar whether or not it was considered to be related to the [18F]FLT.

**Adverse Reaction:** An **Adverse Reaction** is any adverse event caused by a drug. In this study the drug is [<sup>18</sup>F]FLT.

**Suspected adverse reaction** means any adverse event for which there is a reasonable possibility that the drug caused the adverse event. For the purposes of IND safety reporting, "reasonable possibility" means there is evidence to suggest a causal relationship between the drug and the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than adverse reaction, which means any adverse event caused by a drug.

An adverse event or suspected adverse reaction is considered "unexpected" if it is not listed in the investigator brochure or is not listed at the specificity or severity that has been observed; or, if an investigator brochure is not required or available, is not consistent with the risk information described in the general investigational plan or elsewhere in the current application.

An adverse event or suspected adverse reaction is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes: Death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events

include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.

An adverse event or suspected adverse reaction is considered "life-threatening" if, in the view of either the investigator or sponsor, its occurrence places the patient or subject at immediate risk of death. It does not include an adverse event or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

**Investigational Agent:** An investigational agent is any agent held under an Investigational New Drug (IND) application. For purposes of this study, 3'-deoxy-3'-[<sup>18</sup>F]-fluorothymidine ([<sup>18</sup>F]FLT) is the investigational agent.

### 6.iii.8.b. AE Reporting Requirements

The investigators on this protocol will report any suspected adverse events that occur after [18F]FLT administration and within the specified follow-up period to the sponsor, J. Link, and they will work together to determine whether there was an adverse event or adverse reaction and the severity of the adverse event or reaction.

All AEs will be followed by the investigators until resolution, stabilization, scientifically and clinically satisfactory explanation as to attribution and etiology is achieved, or until subject is lost to follow up.

### 6.iii.8.c. CAEPR / ASAE for 3'-deoxy-3'-[18F]fluorothymidine. (NSC 743144)

The Comprehensive Adverse Event and Potential Risks list (CAEPR) provides a single list of reported and/or potential adverse events (AE) associated with an agent using a uniform presentation of events by body system. The Agent Specific Adverse Event List (ASAEL) would include the expected adverse events associated with the use of [18F]FLT. At this time there have been no reported AEs associated with the use of [18F]FLT and so no ASAE are expected as a result of IV injection of [18F]FLT in our study population with the specifications for our drug product (Section 7 of this IND). We will continue to update our CAEPR and ASAE lists as this study progresses, including by reviewing the literature and our in-house data safety monitoring. If any are found we will begin a ASAE list. Any information on reported AEs for [18F]FLT will be provided by the sponsor to all of the investigators on this protocol.

### 6.iii.8.d. Potential but Unexpected Adverse Events for [18F]FLT

The following are extremely rare potential risks that are associated with the use of IV injected radiopharmaceuticals that could apply to the IV administration of I<sup>18</sup>FIFLT.

There is the potential with intravenous injections, including [<sup>18</sup>F]FLT, for allergic reactions and potentially anaphylaxis. This would be a serious to life threatening adverse event. This has not been observed in limited human

exposure to date. Throughout the PET procedure, patients will be monitored by trained personnel for any symptoms or signs of an allergic reaction. Emergency equipment and medical personnel are available in the event of an allergic reaction.

The injection site may become infected.

The dose might be extravasated leading to localized pain / discomfort.

3'-Deoxy-3'-[18F]fluorothymidine is a positron emitting radiopharmaceutical. As such, it poses an intrinsic radiation exposure risk. However, when administered in accordance with the Investigator's Brochure as a PET imaging agent, this risk is felt to be extremely small. The organ and total body doses associated with FLT PET imaging are comparable to those associated with other widely used clinical nuclear medicine procedures and are presented in Section 10 of this IND application.

**Note**: Although not previously reported, in combination with other agents, it is possible that [18F]FLT could exacerbate an adverse event currently known to be caused by an other agent, or might result in adverse events that have not previously been associated with either agent.

### 6.iii.8.e. Review of Safety Information.

As required by 21 CFR 312.32(b), the sponsor will promptly review all information relevant to the safety of the drug. This work will in all cases be done in close collaboration with the physician investigators for this protocol. The physician investigators will be providing much of this information to the local IRB as well for data safety and review monitoring. The sponsor's review will include determining whether there is a safety event over time and the causality. As there are no expected events all events that will be monitored will be unexpected. Reporting will be as described in Table 6.iii.1.

Characterization of the severity of an Adverse Event: Adverse events will be graded as below and based on the definitions in section 6.iii.8.1.

**Grade:** Grade denotes the **severity** of the AE. An AE is graded using the following categories:

- Mild
- Moderate
- Severe
- Life-threatening or disabling
- Fatal

**NOTE**: Severity is graded on the Cancer Therapy Evaluation Program (CTEP) Common Terminology Criteria for Adverse Events (CTCAE) based scale for each adverse event. For example, an abnormal hemoglobin value is graded for severity from 1 to 5 [death] based upon where that value falls on the CTCAE scale of abnormal hemoglobin values. "Severity" is NOT the same as

"Seriousness." All appropriate clinical areas should have access to a copy of the most current CTCAE and a copy of the CTCAE can be downloaded from (http://ctep.cancer.gov).

**Attribution of cause:** The physician investigators will determine whether an adverse event was related to a medical treatment or procedure. Definitions taken from our work with CTEP and NIH give the following definitions for "Attribution" that we will adopt for this IND study: Attribution is a clinical determination, by the investigator, as to whether an AE is related to a medical treatment or procedure. Attribution categories are:

- Definite: The AE is clearly related to a treatment or procedure
- Probable: The AE is likely related to a treatment or procedure
- Possible: The AE may be related to a treatment or procedure
- Unlikely: The AE is likely unrelated to a treatment or procedure
- Unrelated: The AE is clearly not related to a treatment or procedure

**NOTE:** Attribution is part of the assessment of an adverse event. Determining that an event is 'unlikely related' or 'unrelated' to a study agent or procedure does NOT make the event unreportable, or disqualify the event as an AE. As defined above, an AE is reportable as specified herein if it occurred: "during the Adverse Event reporting period defined in the protocol, or by applicable guidance, regulation, or policy."

### 6.iii.8.f. Adverse Event Reporting

Expedited AE reporting for this study will be done through the Cancer Consortium IRB and FDA and as required by FDA MedWatch. These requirements are briefly outlined in the table below.


Table 6.iii.2 Reporting Requirements

| | Unexpected | | | Expected |
|---|---|---|---|---|
| | Adverse Reaction (known or suspected attributable to the use of [18F]FLT) | | AE not<br>attributable to<br>[ <sup>18</sup> F]FLT | AE, AR |
| Reporting<br>Time<br>Requirement<br>to the FDA | Serious including life-threatening (or death) Report to FDA ASAP and within 7 days of discovery of event (section | Annual Continuation Review submission | Life-Threatening or<br>serious or not<br>serious<br>Annual Continuation<br>Review submission | Not<br>applicable to<br>[18F]FLT<br>Not<br>applicable to<br>[18F]FLT |
| Reporting<br>Form for the<br>FDA | 6.iii.8.7) IND Safety report of potentially serious risk | Annual Reports / Case reports | Annual Reports /<br>Case reports | Not<br>applicable to<br>[18F]FLT |
| Reporting<br>Time<br>Requirement<br>to the local<br>IRB | Report to IRB ASAP within 10 days of discovery of event (suspected is defined as 50% probability attributable to [18F]FLT study) this also includes any increased risks with the study even without an AE | At continuation review time | At continuation review time | Not<br>applicable to<br>[ <sup>18</sup> F]FLT |
| Reporting<br>form for the<br>IRB | Expedited Reporting<br>Form for<br>Unanticipated<br>Problems or<br>Noncompliance and<br>Adverse Event<br>Reporting Form | Form for Unanticipated Problems or Noncompliance, Case reports on continuation form, Data Safety Monitoring Reports | Form for<br>Unanticipated<br>Problems or<br>Noncompliance,<br>Case reports on<br>continuation form,<br>Data Safety<br>Monitoring Reports | Not<br>applicable<br>to [18F]FLT |

### 6.iii.8.g. Expedited Adverse Reaction Reporting Guidelines

Life-threatening (or fatal) adverse reactions must be reported within 7 days to the FDA. The FDA should be notified as soon as the adverse reaction is discovered by telephone or fax or email. The instructions and forms are available at <a href="http://www.fda.gov/Safety/MedWatch/HowToReport/default.htm">http://www.fda.gov/Safety/MedWatch/HowToReport/default.htm</a> The report should be sent ASAP by mail and followed with a follow-up report. Individual IND safety reports to FDA are submitted on the Medwatch FDA Form 3500A as an "IND Safety Report". The form should be sent to The Director, Office of Generic Drugs in the Center for Drug Evaluation and Research at FDA. The address and phone numbers are available at: <a href="http://www.fda.gov/AboutFDA/CentersOffices/CDER/ucm119100.htm">http://www.fda.gov/AboutFDA/CentersOffices/CDER/ucm119100.htm</a>.

All life threatening adverse reactions reports are submitted to the FDA, our local IRB and to all investigators. A copy of the report is kept on file.

### 6.iii.8.h. Protocol-Specific Expedited Adverse Event Reporting Exclusion

Not applicable for this IND agent

### 6.iii.8.i. Routine Adverse Event Reporting

Routine Adverse Event Reporting will be done to both the FDA and local IRB as detailed in the table 6.iii.2

### 6.iii.9. PHARMACEUTICAL INFORMATION

### 6.iii.9.a. Production of the Radiopharmaceutical

**3'-Deoxy-3'-**[<sup>18</sup>**F]fluorothymidine (FLT)**: will be produced at the University of Washington according to the methods described in Section 7 of this IND (Chemistry, Manufacturing and Controls).

### 6.iii.9.b. Reported Adverse Events and Potential Risks

A list of the adverse events and potential risks associated with [18F]FLT are provided in Section 6.iii.8.

### 6.iii.9.c. Agent Accountability

The chemical precursor for [18F]FLT is provided by ABX in single-use, 10 mg vials that are delivered to the custody of Dr. Steven Shoner, the lead radiochemist for this project. They are stored in a controlled temperature refrigerator in a locked and secure room and they are inventoried with a chain of custody maintained from the time of receipt. Each radiosynthesis is done by Dr. Shoner, Dr. Krohn or their designee and, after passing all required quality control assays, the product [18F]FLT dose is drawn up under the authority of the nuclear medicine physician co-investigator, Dr. Andrew Shields, Dr. Jean Lee or their designee. The quality control tests that must be passed prior to release of the product [18F]FLT for injection include the pH, radioactive purity, radiochemical purity, specific activity, sterilizing filter integrity, tests for Kryptofix [2.2.2], acetonitrile, acetone, dimethylsulfoxide, endotoxins and particulates. Acceptance criteria are detailed in the CMC section of this IND. The [18F]FLT dose is drawn up into a syringe, assayed for mCi at time of injection, labeled and passed to the physician investigator who oversees the re-assay of the dose and the administration to the research subject.


### 6.iii.10. CORRELATIVE / SPECIAL STUDIES

Study data are comprised of imaging parameters from at least two and as many as four [18F]FLT PET studies.

### 6.iii.10.a. [18F]FLT PET/CT Image Analysis

Preliminary data suggests that [ $^{18}$ F]FLT is essentially irreversibly phosphorylated and trapped inside cells during the imaging period. Prior to this point, however, there is a flux of unphosphorylated [ $^{18}$ F]FLT (reversible component). If the rate of phosphorylation ( $k_3$ ) is low, then the early contribution of perfusion to the measured tumor activity is high. Assuming the phosphorylation rate correlates to the proliferative rate, a high rate of phosphorylation means that the cumulative measured tumor activity should be representative of cellular proliferation.

Volumes of interest (VOIs) will be drawn around the target lesions on the [18F]FLT images based on the tumor localization on the baseline CT. [18F]FLT PET studies will be registered based on their corresponding CT transmission scans images, and time activity curves (TACs) will be calculated.



**Figure 6.iii.3** Kinetic model of FLT metabolism is comprised of an exchangeable tissue compartment and a compartment of trapped FLT \ nucleotides. Four rate constants describe kinetic transfer rates between the 2 compartments. FLTMP = FLT-monophosphate; FLTDP = FLT-diphosphate; FLTTP = FLT-triphosphate; FLT-gluc = FLT-glucuronide;  $Q_e$  = exchangeable tissue compartment;  $Q_m$  = compartment of trapped FLT phosphorylated nucleotides;  $C_{pFLT}$  = concentration of FLT in arterial plasma;  $C_{met}$  = concentration of metabolites in arterial plasma. An imaged extraction procedure will be used to recover the arterial input function (O'Sullivan, et al. 2010).

### 6.iii.10.a.1. Compartmental Analysis

From PET/CT VOI analysis of dynamic data, SUV (30-60 min summed) and parameters reflecting transport ( $K_1$ ) and FLT flux ( $K_{\text{FLT}}$ ) will be calculated using mathematical modeling analysis as described by Muzi et al (Muzi, 2005a; Muzi, 2005b). The change in these rate parameters between baseline and follow up imaging will also be calculated.

### 6.iii.10.b. Biologic Correlates

### **Blood Collection Time Points**

Blood samples will be obtained from each participant at the time of dynamic PET imaging. Each blood sample is used both for the determination of radioactivity and metabolite analysis. Blood samples are drawn from patients using a second venous catheter placed in the opposite arm from the injection site or from a clinically placed PICC line or Port-a-cath. Blood samples of 2-3 mL each are collected into heparinized syringes (or a heparinized blood vacutainer) at 15, 30 and 60 minutes after <sup>18</sup>F-FLT injection, which is infused over one minute

No tissue sampling other than what is required for clinical diagnosis will be done for this study. At the time of resection (or re-resection), tissue not needed for standard clinical care may be labeled with anatomic location co-registered to the PET images and banked for potential future analysis of biomarkers. Any biomarker studies would be described in a separate IRB protocol and would be consented separately from the FLT PET/CT imaging protocol. This consent is already part of the consent for surgery.

### 6.iii.11. STUDY CALENDAR

Table 6.iii.4

| | Pre-<br>Study | Day of [18F]FLT baseline | Mid-Rx | Post-therapy<br>Day of<br>[ <sup>18</sup> F]FLT<br>(optional) | Post-Rx 1 year or time of suspected recurrence [18F]FLT |
|---|---|---|---|---|---|
| Confirmed diagnosis of malignant brain tumor | Х | | | | |
| Informed Consent | Х | - 20 | | | |
| Demographics | Х | | | | |
| Pregnancy Test ** | | Х | | X | X |
| Vital Signs * | х | | | | |
| [ <sup>18</sup> F]FLT Injection and<br>Blood Collection | | х | х | х | х |
| Adverse Event<br>Evaluation | | X (0-24hr) | X (0-24hr) | X (0-24hr) | X (0-24hr) |

<sup>\*</sup>Vital signs include heart rate and blood pressure. \*\* Females of childbearing potential will have a serum pregnancy test just prior to the first PET scan

### 6.iii.12. MEASUREMENT OF EFFECT

This protocol is limited to developing relationships between parameters determined from imaging studies and clinical outcome, which includes treatment assessment using clinical MRI scans. The definition of response is defined below using Tables 6.iii.5 and 6.iii.6 from Wen et al., (Wen 2010). The RANO criteria do not rely on two

dimensional volume assessments in the MRI image for determination of response status.

**Table 6.iii.5.** Criteria for Response Assessment Incorporating MRI and Clinical Factors (Wen 2010)

| Response | Criteria |
|---|---|
| Complete<br>response | Requires all of the following: complete disappearance of all enhancing measurable and nonmeasurable disease sustained for at least 4 weeks; no new lesions; stable or improved nonenhancing [T2/FLAIR] lesions; patients must be off corticosteroids [or on physiologic replacement doses only], and stable or improved clinically. Note: Patients with nonmeasurable disease only cannot have a complete response; the best response possible is stable disease. |
| Partial<br>response | Requires all of the following: >50% decrease compared with baseline in the sum of products of perpendicular diameters of all measureable enhancing lesions sustained for at least 4 weeks; no progression or nonmeasurable disease; no new lesions; stable or improved nonenhancing [T2/FLAIR] lesions on same or lower dose of corticosteroids compared with baseline scan; the corticosteroid dose at the time of the scan evaluation should be no greater than the dose at time of baseline scan, and stable or improved clinically. Note: Patients with nonmeasurable disease only cannot have a partial response; the best response possible is stable disease. |
| Stable<br>disease | Requires all of the following: does not qualify for complete response, partial response, or progression; stable nonenhancing [T2/FLAIR] lesions on same or lower dose of corticosteroids compared with baseline scan. In the event that the corticosteroid doses was increased for new symptoms and signs without confirmation of disease progression on neuroimaging, and subsequent follow-up imaging shows that the increase in corticosteroids was required because of disease progression, the last scan considered to show stable disease will be the scan obtained when the corticosteroid dose was equivalent to the baseline dose. |
| Progression | Defined by any of the following: ≥25% increase in sum of the products of perpendicular diameters of enhancing lesions compared with the smallest tumor measurement obtained either at baseline (or no decrease) or best response, one stable or increasing doses of corticosteroids*; significant increase in T2/FLAIR nonenhancing lesion on stable or increasing doses of corticosteroids compared with baseline scan or best response after initiation of therapy* not caused by comorbid events (e.g. radiation therapy, demyelination, ischemic injury, infection, seizures, postoperative changes, or other treatment effects); any new lesion; clear clinical deterioration not attributable to other causes apart from the tumor (e.g. seizures, medication adverse effects, complications of therapy, cerebrovascular events, infection, and so on) or changes in corticosteroid dose; failure to return for evaluation as a result of death or deteriorating condition; or clear progression of nonmeasurable disease. |
| technique as at base Abbreviations: MRI, | le and nonmeasurable lesions must be assessed using the same |
| recovery. *Stable doses of cort | icosteroids include patients not on corticosteroids. |

Table 6.iii.6 Summary of the Proposed RANO Response Criteria

| Criterion | CR | PR | SD | PD |
|---|---|---|---|---|
| T1 gadolnium<br>enhancing<br>disease | None | ≥ 50% ♥ | < 50% <b>√</b> but <25% <b>↑</b> | ≥ 25% ↑* |
| T2/FLAIR | Stable or <b>Ψ</b> | Stable or <b>Ψ</b> | Stable or <b>Ψ</b> | ↑* |
| New lesion | None | None | None | Present* |
| Corticosteroids | None | Stable or <b>Ψ</b> | Stable or <b>Ψ</b> | NA <sup>Δ</sup> |
| Clinical Status | Stable 1 | Stable or 1 | Stable or 1 | Ψ* |
| Requirement for response | All | All | All | Any* |

Abbreviations: RANO, Response Assesement in Neuro-Oncology; CR, complete response; PR, partial response; SD, stable disease; PD, progressive disease; FLAIR, fluid-attenuated inversion recover; NA, not applicable

The primary analysis variables for the study are:

- Percentage change in K<sub>1</sub>, FLT flux and SUV for [<sup>18</sup>F]FLT PET/CT
- Assessment of clinical response per the response criteria listed above.
- Survival

Secondary analysis variables are:

- Heterogeneity in K<sub>1</sub>, FLT flux and SUV for [<sup>18</sup>F]FLT PET/CT at baseline
- Comparison of heterogeneity at different times

### 6.iii.13. DATA REPORTING / REGULATORY CONSIDERATIONS

Adverse event lists, guidelines, and instructions for AE reporting are described in Section 6.iii.8. The Principal Physician Investigator is responsible for maintaining complete and timely, HIPAA-compliant electronic records of clinical and image datasets.

### 6.iii.14. STATISTICAL CONSIDERATIONS

### 6.iii.14.a. Study Description

This is a study involving [<sup>18</sup>F]FLT PET/CT imaging of patients with brain tumors at different times during the course of standard treatment. Thirty patients with brain tumors and who are planning standard therapy with surgical resection, chemotherapy or radiotherapy or any combination, will be enrolled. We will evaluate the values for percentage changes in [<sup>18</sup>F]FLT PET measures observed following 1-3 weeks of therapy, shortly after finishing therapy and at time of

<sup>\*</sup> Progression occurs when this criterion is present.

 $<sup>\</sup>Delta$  Increase in corticosteroids alone will not be taken into account in determining progression in the absence of persistent clinical deterioration.

recurrence or at one year, which ever comes first and explore associations between [18F]FLT PET parameters and their changes and clinical outcome.

### 6.iii.14.b. Power Calculations

For hypotheses 2 and 3, we will use patient survival as our outcome variable and the analysis will be based on the Cox proportional hazards model with adjustment for confounding. We have estimated that with 30 patients our study will have power characteristics presented in Table 6.iii.7. These calculations used a value for the study effect of 0.75.

| Table 6.iii.7. Power calculation for measuring response | FU=2 yrs | FU=7 yrs |
|---|---|---|
| Power without cofounders | 0.79 | 0.80 |
| Power using cofounders, including FDG PET/CT | 0.87 | 0.83 |
| Effect of 15% measurement error | 0.89 | 0.84 |

The analysis of data for these hypotheses involves within-subject changes where the variance in values will be less than between-subject FLT results that we have published. Furthermore, this power analysis has assumed that only data from a single volume of interest (VOI) for each subject will be used. In the context of our aims, this could be considered inefficient. In many subjects it will be possible to include data from spatially well-separated and hence substantially uncorrelated sub-regions within large tumors (Spence,1998) as distinct sampling units for consideration with this hypothesis. Not withstanding the additional variability that sub-region measurements will have, it is likely that some gains in statistical precision can be realized by this approach. Thus the 90% power estimate is conservative.

Hypothesis 1. Among GBM patients identified as progressing according to Macdonald criteria at 1-month follow-up, the mean FLT flux in true progression cases will be compared to the corresponding mean in the pseudo-progression cases. Preliminary data indicate that 40% of MRI diagnosed progression can be expected to be pseudo-progression. Our data on recurrence vs radionecrosis for KFLT recurrences showed a mean of 0.017 and a standard deviation of 0.005 (Spence, 2006). The mean of the radionecrosis group was 0.004, roughly one-quarter for that for recurrences. Thus, conservatively, assuming that pseudo-progressors showed even a 30% increase over the mean KFLT value, the expected difference between the groups would be 0.017x0.3 or about 0.005. From this, the expected standardized effect is 0.99. Using a 2-sample t-test with significance level of 5% for assessment of the hypothesis, the power of our study is about 95%

### 6.iii.14.c. Analysis Plan

Percentage change between pre-treatment and post-therapy measurements will be computed for [18F]FLT PET/CT measures of transport, K1, and flux (KFLT). Log transformations will be considered if the rates of change are highly skewed. Outcome analysis studies are directed toward predicting tumor response. In the case of progression, a multivariate logistic regression will be used to produce an analysis of how the combination of standard diagnostics plus the FLT parameters (K1, KFLT, SUVmean) obtained shortly after therapy can best be combined to

obtain a prognostic variable for determination of progression. Although the prognostic variable will provide a direct assessment of the probability of response for an individual patient, we will also develop a ROC characterization of its diagnostic performance. We fully appreciate that the small number of patients means that this analysis may suffer from a lack of power but it should be useful in planning a larger follow-up if the results are encouraging.

A similar approach will be used for survival analysis.. Here we will use multivariate Cox regression analysis with both baseline and follow-up variables to be considered.

The heterogeneity of the within-tumor proliferation obtained by application of the elliptical heterogeneity measure developed by Eary et al (2008) will be used in a secondary analysis.

### 6.iii.14.d. Stratification Factors

Not Applicable.

### 6.iii.14.e. Reporting and Exclusions

Evaluation of Toxicity: All patients will be evaluable for toxicity from their [18F]FLT PET.

### 6.iii.15. LITERATURE CITED

Bibikova M, Yeakley JM, Wang-Rodriguez J, Fan JB. Quantitative expression profiling of RNA from formalin-fixed paraffin-embedded tissues using randomly assembled bead arrays. *Methods Mol Biol* 2008; *439* 159-77.

Brandes AA, Franceschi E, Tosoni A, Blatt V, Pession A, Tallini G, Bertorelle R, Bartolini S, Calbucci F, Andreoli A, Frezza G, Leonardi M, Spagnolli F, Ermani M. MGMT promoter methylation status can predict the incidence and outcome of pseudoprogression after concomitant radiochemotherapy in newly diagnosed glioblastoma patients. *J Clin Oncol*. 2008 May 1; 26(13) 2192-7.

Buckner JC, Ingle JN, Everson LK, O'Fallon JR, Cullinan SA, Ahmann DL, Krook JE, Pfeifle DM. Results of salvage hormonal therapy and salvage chemotherapy in women failing adjuvant chemotherapy after mastectomy for breast cancer. *Breast Cancer Res Treat* 1989; *13* (2) 135-42.

Carlson RW. Sequencing of endocrine therapies in breast cancer--integration of recent data. *Breast Cancer Res Treat* 2002; 75 Suppl 1 S27-32; discussion S33-5.

Carlson RW, McCormick B. Update: NCCN breast cancer Clinical Practice Guidelines. *J Natl Compr Canc Netw* 2005; 3 Suppl 1 S7-11.

Carlson RW, Allred DC, Anderson BO, Burstein HJ, Carter WB, Edge SB, Erban JK, Farrar WB, Goldstein LJ, Gradishar WJ, Hayes DF, Hudis CA, Jahanzeb M, Kiel K,

Ljung BM, Marcom PK, Mayer IA, McCormick B, Nabell LM, Pierce LJ, Reed EC, Smith ML, Somlo G, Theriault RL, Topham NS, Ward JH, Winer EP, Wolff AC. Breast cancer. Clinical practice guidelines in oncology. *J Natl Compr Canc Netw* 2009; 7 (2) 122-92.

Chen W, Cloughesy T, Kamdar N, Satyamurthy N, Bergsneider M, Liau L, Mischel P, Czernin J, Phelps ME, Silverman DH. Imaging proliferation in brain tumors with <sup>18</sup>F-FLT PET: comparison with <sup>18</sup>F-FDG. *J Nucl Med* 2005; *46* (6) 945-52.

Chia SK, Speers CH, D'Yachkova Y, Kang A, Malfair-Taylor S, Barnett J, Coldman A, Gelmon KA, O'Reilly SE, Olivotto IA. The impact of new chemotherapeutic and hormone agents on survival in a population-based cohort of women with metastatic breast cancer. *Cancer* 2007; *110* (5) 973-9.

de Wit MC, de Bruin HG, Eijkenboom W, Sillevis Smitt PA, van den Bent MJ. Immediate post-radiotherapy changes in malignant glioma can mimic tumor progression. *Neurology*. 2004 Aug 10;63(3):535-7.

Dowsett M, Smith IE, Ebbs SR, Dixon JM, Skene A, Griffith C, Boeddinghaus I, Salter J, Detre S, Hills M, Ashley S, Francis S, Walsh G. Short-term changes in Ki-67 during neoadjuvant treatment of primary breast cancer with anastrozole or tamoxifen alone or combined correlate with recurrence-free survival. *Clin Cancer Res* 2005; *11* (2 Pt 2) 951s-8s.

Dowsett M, Smith IE, Ebbs SR, Dixon JM, Skene A, A'Hern R, Salter J, Detre S, Hills M, Walsh G. Prognostic value of Ki67 expression after short-term presurgical endocrine therapy for primary breast cancer. *J Natl Cancer Inst* 2007; 99 (2) 167-70.

Early Breast Cancer Trials Group. Tamoxifen for early breast cancer: an overview of the randomised trials. Early Breast Cancer Trialists' Collaborative Group. *Lancet* 1998; 351 (9114) 1451-67.

Ellis MJ. Improving outcomes for patients with hormone receptor-positive breast cancer: back to the drawing board. *J Natl Cancer Inst* 2008; *100* (3) 159-61.

Eriksson S, Arnér E, Spasokoukotskaja T, Wang L, Karlsson A, Brosjö O, Gunvén P, Julusson G, Liliemark J. Properties and levels of deoxynucleoside kinases in normal and tumor cells; implications for chemotherapy. *Adv Enzyme Regul*. 1994;34:13-25.

Fabrini MG, Perrone F, De Franco L, Pasqualetti F, Grespi S, Vannozzi R, Cionini L. Perioperative high-dose-rate brachytherapy in the treatment of recurrent malignant gliomas. *Strahlenther Onkol.* 2009 Aug;185(8):524-9.

Fokas E, Wacker U, Gross MW, Henzel M, Encheva E, Engenhart-Cabillic R. Hypofractionated stereotactic reirradiation of recurrent glioblastomas: a beneficial treatment option after high-dose radiotherapy? *Strahlenther Onkol*. 2009 Apr;185(4):235-40.

Greenberg PA, Hortobagyi GN, Smith TL, Ziegler LD, Frye DK, Buzdar AU. Long-term follow-up of patients with complete remission following combination chemotherapy for metastatic breast cancer. *J Clin Oncol* 1996; *14* (8) 2197-205.

Jemal A, Siegel R, Ward E, Murray T, Xu J, Smigal C, Thun MJ. Cancer statistics 2006. *CA Cancer J Clin* 2006; *56* (2) 106-30.

Jemal A, Ward E, Thun MJ. Recent trends in breast cancer incidence rates by age and tumor characteristics among U.S. women. *Breast Cancer Res.* 2007; 9(3): R28.

Jemal A, Siegel R, Xu J, Ward E. Cancer statistics 2010. CA Cancer J Clin 60 (5) 277-300.

Kenny L Coombes RC, Vigushin DM, Al-Nahhas A, Shousha S, Aboagye EO. Imaging early changes in proliferation at 1 week post chemotherapy: a pilot study in breast cancer patients with 3'-deoxy-3'-[18F]fluorothymidine positron emission tomography. *Eur J Nucl Med Mol Imaging* 2007; *34* (9) 1339-47

Krohn KA and Grierson J R, Muzi M, and Schwartz JL, "Radiopharmaceuticals for Imaging Proliferation," in Targeted Molecular Imaging, eds. M. J. Welch and W. C. Eckelman. Boca Raton, FL: CRC Press 2012, pp. 231-251.

Lancaster HO. Significance tests in discrete distributions. *Journal of the American Statistical Association* 1961; *56* 223-234.

Leyton J, Latigo JR, Perumal M, Dhaliwal H, He Q, Aboagye EO. Early detection of tumor response to chemotherapy by 3'-deoxy-3'-[18F]fluorothymidine positron emission tomography: the effect of cisplatin on a fibrosarcoma tumor model in vivo. *Cancer Res* 2005; 65 (10) 4202-10.

Li Cl, Daling JR, and Malone KE. Incidence of invasive breast cancer by hormone receptor status from 1992 to 1998. *J Clin Oncol*. 2003; 21(1): 28-34.

Lonning PE, Taylor PD, Anker G, Iddon J, Wie L, Jorgensen LM, Mella O, Howell A. High-dose estrogen treatment in postmenopausal breast cancer patients heavily exposed to endocrine therapy. *Breast Cancer Res Treat* 2001; 67 (2) 111-6.

Mouridsen H, Gershanovich M, Sun Y, Perez-Carrion R, Boni C, Monnier A, Apffelstaedt J, Smith R, Sleeboom HP, Janicke F, Pluzanska A, Dank M, Becquart D, Bapsy PP, Salminen E, Snyder R, Lassus M, Verbeek JA, Staffler B. Chaudri-Ross HA. Dugan M. Superior efficacy of letrozole versus tamoxifen as first-line therapy for postmenopausal women with advanced breast cancer: results of a phase III study of the International Letrozole Breast Cancer Group. *J Clin Oncol* 2001; *19* (10) 2596-606.

Muzi M, Spence AM, O'Sullivan F, Mankoff DA, Wells MW, Grierson JR, Link JM, Krohn KA. Kinetic analysis of 3'-deoxy-3'-18F- flourothymidine in patients with gliomas. *J Nucl Med.* 2006; 47(10):1612-21.

Muzi M, Vesselle H. Kinetic analysis of 3'-deoxy-3'-fluorothymidine PET studies: validation studies in patients with lung cancer. *J Nucl Med.* 2005a; 46(2):274-82.

Muzi M, Mankoff DA, Grierson JR, Wells JM, Vesselle H, Krohn K,A. Kinetic modeling of 3'-deoxy-3'-fluorothymidine in somatic tumors: mathematical studies. *J Nucl Med* 2005b; 46 (2) 371-80.

Nabholtz JM, Buzdar A, Pollak M, Harwin W, Burton G, Mangalik A, Steinberg M, Webster A, von Euler M. Anastrozole is superior to tamoxifen as first-line therapy for advanced breast cancer in postmenopausal women: results of a North American multicenter randomized trial. Arimidex Study Group. *J Clin Oncol* 2000; 18 (22) 3758-67.

Osborne CK. Tamoxifen in the treatment of breast cancer. *N Engl J Med* 1998 339 (22) 1609-18.

Osborne CK, Pippen J, Jones SE, Parker LM, Ellis M, Come S, Gertler SZ, May JT, Burton G, Dimery I, Webster A, Morris C, Elledge R, Buzdar A. Double-blind randomized trial comparing the efficacy and tolerability of fulvestrant versus anastrozole in postmenopausal women with advanced breast cancer progressing on prior endocrine therapy: results of a North American trial. *J Clin Oncol* 2002; 20 (16) 3386-95.

O'Sullivan F, Kirrane J, Muzi M, O'Sullivan JN, Spence AM, Mankoff DA, Krohn KA. (2010) Kinetic quantitation of cerebral PET-FDG studies without concurrent blood sampling: statistical recovery of the arterial input function. *IEEE Trans Med Imaging*. 29(3):610-624.

Piccart-Gebhart MJ. Moving away from the "one shoe fits all" strategy: the key to future progress in chemotherapy. *J Clin Oncol* 2005; 23 (8) 1611-3.

Romond EH, Perez EA, Bryant J, Suman VJ, Geyer CE, Jr, Davidson NE, Tan-Chiu E, Martino S, Paik S, Kaufman PA, Swain SM, Pisansky TM, Fehrenbacher L, Kutteh LA, Vogel V G, Visscher DW, Yothers G, Jenkins RB, Brown AM, Dakhil SR, Mamounas EP, Lingle W, L, Klein PM, Ingle JN, Wolmark N. Trastuzumab plus adjuvant chemotherapy for operable HER2-positive breast cancer. *N Engl J Med* 2005; *353* (16) 1673-84.

Sathornsumetee S, Reardon DA. Targeting multiple kinases in glioblastoma multiforme. *Expert Opin Investig Drugs*. 2009 Mar;18(3):277-92.

Schwartz JL, Tamura Y, Jordan R, Grierson JR, Krohn K. A. Monitoring tumor cell proliferation by targeting DNA synthetic processes with thymidine and thymidine analogs. *J Nucl Med* 2003; 44 (12) 2027-32.

Shields AF, Grierson JR, Dohmen BM, etc. 1998. Imaging proliferation in vivo with [F-18]FLT and positron emission tomography. *Nat Med* 4(11):1334-6.

Smyczek-Gargya B, Fersis N, Dittmann H, Vogel U, Reischl G, Machulla HJ, Wallwiener D, Bares R, Dohmen BM. PET with [18F]fluorothymidine for imaging of primary breast cancer: a pilot study. *Eur J Nucl Med Mol Imaging* 2004; *31* (5) 720-4.

Storey J D, Tibshirani R. Statistical significance for genomewide studies. *Proc Natl Acad Sci U S A* 2003; *100* (16) 9440-5.

Subramanian A, Tamayo P, Mootha VK, Mukherjee S, Ebert BL, Gillette MA, Paulovich A, Pomeroy SL, Golub TR, Lander E S, Mesirov JP. Gene set enrichment analysis: a knowledge-based approach for interpreting genome-wide expression profiles. *Proc Natl Acad Sci U S A* 2005; *102* (43) 15545-50.

Taal W, Brandsma D, de Bruin HG, Bromberg JE, Swaak-Kragten AT, Smitt PA, van Es CA,

van den Bent MJ. Incidence of early pseudo-progression in a cohort of malignant glioma patients treated with chemoirradiation with temozolomide. *Cancer.* 2008 Jul 15;113(2):405-10.

van Waarde A, Cobben DC, Suurmeijer AJ, Maas B, Vaalburg W, de Vries EF, Jager PL, Hoekstra HJ, Elsinga PH. Selectivity of <sup>18</sup>F-FLT and <sup>18</sup>F-FDG for differentiating tumor from inflammation in a rodent model. *J Nucl Med* 2004; *45* (4) 695-700.

Villano JL, Seery TE, Bressler LR. Temozolomide in malignant gliomas: current use and future targets. *Cancer Chemother Pharmacol*. 2009 Sep;64(4):647-55.

Weber G, Nagai M, Natsumeda Y, Ichikawa S, Nakamura H, Eble JN, Jayaram HN, Zhen WN, Paulik E, Hoffman R, et al. Regulation of de novo and salvage pathways in chemotherapy. *Adv Enzyme Regul*. 1991;31:45-67.

Wells JM, Mankoff DA, Muzi M, et al. 2002a. Kinetic analysis of 2-[11C]thymidine PET imaging studies of malignant brain tumors: compartmental model investigation and mathematical analysis. *Mol Imaging* 1(3):151-59.

Wen PY, Macdonald DR, Reardon DA, Cloughesy TF, Sorenson GA, Galanis G, DeGroot J, Wick W, Glibert MR, Lassman AB, Tsien C, Mikkelsen T, Wong ET, Chamberlain MC, Stupp R, Lamborn KR, Vogelbaum MA, Ven den Bent MJ, Chang SM. Updated response assessment criteria for high grade gliomas: Response Assessment in Neuro-oncology Working Group. *J Clin Oncol* 2010; 28: 1963-1972.

Winer EP, Hudis C, Burstein HJ, Wolff AC, Pritchard KI, Ingle JN, Chlebowski RT, Gelber R, Edge SB, Gralow J, Cobleigh MA, Mamounas EP, Goldstein LJ, Whelan TJ, Powles T J, Bryant J, Perkins C, Perotti J, Braun S, Langer AS, Browman GP. Somerfield M. R. American Society of Clinical Oncology technology assessment on the use of aromatase inhibitors as adjuvant therapy for postmenopausal women with hormone receptor-positive breast cancer: status report 2004. *J Clin Oncol* 2005 23 (3) 619-29.